CLINICAL TRIAL: NCT06791499
Title: AI-Agent Assisted Automation for Diagnosing and Predicting Patients Using Electronic Health Records and Multimodal Data
Brief Title: AI-Agent for Automated Diagnosis and Predicting Using EHR and Multimodal Data
Status: Recruiting | Type: Observational
Sponsor: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Kang Zhang, Chief Scientist, Wenzhou Medical University
Other Study IDs: AI-agent
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: AI Agent
Keywords: AI agent

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AI-Assisted Disease Prediction Using EHR and Imaging Data: This cohort consists of patients whose historical health data, including electronic health records (EHR) and multimodal imaging data (e.g., X-rays, MRIs, CT scans, ultrasounds), will be analyzed by an AI agent. The AI system will assist in diagnosing and predicting diseases by processing and integrating these diverse data sources. The primary focus is to evaluate the ability of the AI agent to identify patterns and predict disease progression with high accuracy. Participants will not be required to take any additional actions beyond providing their medical history and imaging data. The aim is to assess how well the AI system can support clinical decision-making and improve diagnostic outcomes based on the provided data.

SUMMARY:
The goal of this clinical study is to evaluate the effectiveness of an AI agent in diagnosing and predicting diseases using electronic health records (EHR) and multimodal imaging data. The AI agent leverages advanced machine learning algorithms to process and analyze diverse health data sources, aiming to assist healthcare providers in making more accurate diagnoses and predictions.

DETAILED DESCRIPTION:
This multi-center, retrospective clinical study is designed to evaluate the application and effectiveness of an AI agent in the medical decision-making process. The AI agent integrates and analyzes multimodal data, including electronic health records (EHR) and various imaging data (e.g., X-rays, MRIs, CT scans, ultrasounds) to predict and diagnose a range of diseases. By leveraging the power of machine learning and data fusion techniques, the AI agent can identify patterns in large and complex datasets, offering insights that may not be immediately apparent through traditional diagnostic methods.The study will compare the AI agent's diagnostic accuracy and disease prediction capabilities with traditional diagnostic practices to assess its potential benefits in clinical settings. Key questions include whether the AI agent can assist in early diagnosis, predict disease progression, and support healthcare professionals in making personalized treatment decisions. Participants will not be required to undergo any additional interventions; they will only provide historical health data, including EHR and relevant imaging data, which will be analyzed by the AI agent. The AI system will then use this data to assist healthcare providers by offering predictions and diagnostic suggestions based on the analysis of the multimodal information. The ultimate goal is to determine whether this AI-driven approach can improve diagnostic accuracy, optimize treatment strategies, and enhance patient outcomes in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have comprehensive electronic health records (EHR) available, including demographic information, medical history, and laboratory results.
2. Participants must have available multimodal imaging data (e.g., X-rays, CT scans, MRIs, ultrasounds) relevant to their health condition.
3. Participants must have a confirmed diagnosis of one or more diseases or health conditions based on clinical records or imaging data.
4. Patients must provide consent for the use of their historical health data for research purposes.

Exclusion Criteria:

1. Participants with ambiguous or unverifiable diagnoses that cannot be accurately categorized.
2. Duplicate or redundant patient data (e.g., repeated records of the same patient without clear differentiation).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participants for this study will be selected from multiple healthcare centers and hospitals that maintain comprehensive electronic health records (EHR) and multimodal imaging data. The study population will include patients who have a variety of diseases or health conditions, with data available for diagnosis and disease progression. Participants will have confirmed diagnoses based on clinical records or imaging data, including but not limited to conditions captured by X-rays, CT scans, MRIs, and ultrasounds. Both those with complex health conditions and those with more common illnesses will be included to evaluate the AI system's diagnostic and predictive capabilities across a broad spectrum of cases.Participants from these centers will provide historical health data, and there will be no active intervention beyond the use of their existing clinical and imaging data for training and testing the AI system.
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | 1 year
  AUC of the ROC curve, used to quantify diagnostic accuracy. No unit (a ratio or percentage, typically expressed as a number between 0 and 1).
F1 Score | 1 year
  The F1 score is the harmonic mean of precision and sensitivity (recall). It is a good measure of the model's ability to identify both true positives and minimize false positives, especially in cases where the classes are imbalanced (e.g., when the number of healthy cases is much higher than disease cases). The F1 score ranges from 0 to 1, with 1 indicating perfect precision and recall.

SECONDARY OUTCOMES:
Sensitivity (True Positive Rate) | 1 year
  Sensitivity measures how well the AI model identifies true positive cases, such as correctly diagnosing pregnant women with complications or identifying neonatal disorders.
Specificity (True Negative Rate) | 1 year
  Specificity measures the ability of the AI model to correctly identify cases without diseases, ensuring that healthy mothers and infants are correctly identified as negative.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Hospital, Guangzhou, Guangdong
  - West China Hospital, Chengdu, Sichuan
  - First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No